CLINICAL TRIAL: NCT00660985
Title: A Pharmacokinetic Study to Compare the Systemic Exposure to Adapalene During Dermal Application of Either Differin® Gel, 0.3% (Adapalene 0.3%) or Differin® Gel, 0.1% (Adapalene 0.1%) for 30 Days in Subjects With Acne Vulgaris
Brief Title: Pharmacokinetic Study to Compare the Systemic Exposure of Differin® Gel, 0.3% or Differin® Gel, 0.1%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Michael Graeber, MD, Head of US Development:, Galderma R&D
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06.SPR.18115
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Results first posted 2009-12-29 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2011-01

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris; Differin; Adapalene
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Differin® Gel, 0.3% (Experimental): Gel, 0.3%, 2g, once daily for 30 days
  Interventions: Drug: Adapalene
- Differin® Gel, 0.1% (Active Comparator): Gel, 0.1%, 2g, once daily for 30 days
  Interventions: Drug: Adapalene

INTERVENTIONS:
Drug: Adapalene — Gel, 0.3%, 2g, once daily for 30 days
  Arms: Differin® Gel, 0.3%
Drug: Adapalene — Gel, 0.1%, 2g, once daily for 30 days
  Arms: Differin® Gel, 0.1%

SUMMARY:
Phase 4 commitment pharmacokinetic study to determine systemic exposure to adapalene.

DETAILED DESCRIPTION:
Multi-center, double-blind, randomized, parallel group study enrolling male or female subjects with acne vulgaris.

Screening will take place within 14 days prior to Baseline. At the Baseline visit, and at each study day up to Day 30, a trained nurse or technician will apply 2 grams of study medication (either Differin® Gel, 0.3% or Differin® Gel, 0.1%) to the face, upper part of chest, and upper part of back of the subjects. To ensure maximal usage conditions, 2 grams study medication will be applied once daily to a total body surface area of approximately 1000 cm², which is equivalent to 2 mg/cm2.

Subjects will arrive at the clinic the night before on visit days (Day 1, Day 15 and Day 30) when PK blood samples will be drawn. Subjects will be discharged from the clinic on Day 2 and Day 16 following the 24-hour post-dose blood sample, and on Day 31 after the 36-hour post-dose blood samples.

Cutaneous safety (local tolerability assessments) will be assessed, by recording erythema, scaling, dryness, and stinging/burning sensation as separate scores on the face, upper part of the chest, and upper part of the back using a 4-point scale (0 = None to 3 = Severe). Local tolerability assessments will be performed weekly on Day 1, 8, 15, 22 and Day 30, prior application of study medication.

Efficacy will be evaluated by Inflammatory and Non-inflammatory lesion counts on the face performed at Screening, Baseline (Day 1), and on Day 30.

Subjects will have routine laboratory tests (fasting hematology, blood chemistry) performed at Screening and at Day 30 visits.

Blood samples for determination of adapalene plasma concentrations will be drawn on Day 1, Day 15, and Day 30 before the morning study medication application (pre-dose) and 1, 2, 4, 6, 8, 10, 12, 16 and 24 hours after application of study medication; and additionally after the last study medication application (Day 31, 32, 33) at 32, 36, 48 and 72 hours post-dose.

The adapalene plasma concentrations will be determined by a high performance liquid chromatography (HPLC) and fluorescence detection method.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 35 years of age
* Clinical diagnosis of acne vulgaris
* Minimum of 20 Inflammatory
* Minimum of 20 Non-inflammatory lesions
* The subject has a body weight between 45 and 100 kg, and a Body Mass Index (BMI) between 18 and 30Kg/m2

Exclusion Criteria:

* More than 1 nodule or any cyst on the face (excluding the nose)
* Acne conglobata, acne fulminans, secondary acne or severe acne
* Underlying diseases or other dermatological conditions that require the use of interfering topical or systemic therapy
* Pregnant or nursing or planning a pregnancy
* Surgical or medical condition which might interfere with the absorption, distribution, metabolism, or excretion of the drug
* Known allergies to any of the ingredients of the study medication
* History of alcohol or drug abuse or positive test results for any drug abuse
* Positive test results for hepatitis B surface antigen (HBs-Ag), hepatitis C virus (HCV) or human immunodeficiency virus antibodies (HIV Ab)
* Use of prohibited medications prior to the study unless appropriate washout period is documented

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Director — Galderma R&D
Locations (2):
- United States (2):
  - DermResearch, Inc., Austin, Texas
  - J&S Studies, Inc., College Station, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Differin® Gel, 0.3% | Differin® Gel, 0.1%
Started | 26 | 25
Completed | 25 | 25
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Differin® Gel, 0.3% | Differin® Gel, 0.1% | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 25 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.4 (4.87) | 21.3 (3.78) | 22.4 (4.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Cmax (ng/mL) at Day 1
Description: the observed peak drug (adapalene) concentration
Time Frame: T0 (predose), T1hour (hr), T2hr, T4hr, T6 hr, T8 hr, T10hr, T12hr, T16hr, T24hr (post dose)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Differin® Gel, 0.3% | Differin® Gel, 0.1%
Number analyzed (Participants) | 25 | 25
ng/mL | 0.10 (0.10) | 0.02 (0.06)

2. Primary Outcome: Cmax (ng/mL) at Day 15
Description: the observed peak drug (adapalene) concentration
Time Frame: T0 (predose), T1hour (hr), T2hr, T4hr, T6 hr, T8 hr, T10hr, T12hr, T16hr, T24hr (post dose)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Differin® Gel, 0.3% | Differin® Gel, 0.1%
Number analyzed (Participants) | 25 | 25
ng/mL | 0.18 (0.09) | 0.04 (0.08)

3. Primary Outcome: Cmax (ng/mL) at Day 30
Description: the observed peak drug (adapalene) concentration
Time Frame: T0 (predose), T1hour (hr), T2hr, T4hr, T6 hr, T8 hr, T10hr, T12hr, T16hr, T24hr, T32hr, T36hr, T48hr, T 72hr (post dose)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Differin® Gel, 0.3% | Differin® Gel, 0.1%
Number analyzed (Participants) | 25 | 25
ng/mL | 0.15 (0.10) | 0.03 (0.06)

4. Primary Outcome: Tmax (hr) at Day 1
Description: the time at which Cmax occurs
Time Frame: T0 (predose), T1hour (hr), T2hr, T4hr, T6 hr, T8 hr, T10hr, T12hr, T16hr, T24hr (post dose)
Population: 26 subjects in the Differin Gel 0.3% and 25 subjects in the Differin Gel 0.1% were included in the study. 14 subjects in the Differin Gel 0.3% and 4 subjects in the Differin Gel 0.1% were detectable at Day 1.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Differin® Gel, 0.3% | Differin® Gel, 0.1%
Number analyzed (Participants) | 14 | 4
hours | 15 (6) | 11 (4)

5. Primary Outcome: Tmax (hr) at Day 15
Description: the time at which Cmax occurs
Time Frame: T0 (predose), T1hour (hr), T2hr, T4hr, T6 hr, T8 hr, T10hr, T12hr, T16hr, T24hr (post dose)
Population: 26 subjects in the Differin Gel 0.3% and 25 subjects in the Differin Gel 0.1% were included in the study. 23 subjects in the Differin Gel 0.3% and 7 subjects in the Differin Gel 0.1% were detectable at Day 15.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Differin® Gel, 0.3% | Differin® Gel, 0.1%
Number analyzed (Participants) | 23 | 7
hours | 13 (8) | 11 (5)

6. Primary Outcome: Tmax (hr) at Day 30
Description: the time at which Cmax occurs
Time Frame: T0 (predose), T1hour (hr), T2hr, T4hr, T6 hr, T8 hr, T10hr, T12hr, T16hr, T24hr, T32hr, T36hr, T48hr, T72hr (post dose)
Population: 26 subjects in the Differin Gel 0.3% and 25 subjects in the Differin Gel 0.1% were included in the study. 20 subjects in the Differin Gel 0.3% and 4 subjects in the Differin Gel 0.1% were detectable at Day 30.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Differin® Gel, 0.3% | Differin® Gel, 0.1%
Number analyzed (Participants) | 20 | 4
hours | 13 (6) | 12 (3)

7. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve for 0 to 24 Hours Post Dose Measured on Day 1 (AUC (0-24))
Description: area under the concentration-time curve calculated mixed linear-logarithmic trapezoidal method from pre-application (T0) through 24 hr (corresponding to the dosing interval)
Time Frame: T0 (predose), T1hour (hr), T2hr, T4hr, T6 hr, T8 hr, T10hr, T12hr, T16hr, T24hr (post dose)
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Differin® Gel, 0.3% | Differin® Gel, 0.1%
Number analyzed (Participants) | 25 | 25
ng*h/mL | 1.54 (1.58) | 0.31 (0.73)

8. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve for 0 to 24 Hours Post Dose Measured on Day 15 (AUC (0-24))
Description: area under the concentration-time curve calculated mixed linear-logarithmic trapezoidal method from pre-application (T0) through 24hr (corresponding to the dosing interval)
Time Frame: T0 (predose), T1hour (hr), T2hr, T4hr, T6 hr, T8 hr, T10hr, T12hr, T16hr, T24hr (post dose)
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Differin® Gel, 0.3% | Differin® Gel, 0.1%
Number analyzed (Participants) | 24 | 25
ng*h/mL | 2.84 (1.75) | 0.50 (0.99)

9. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve for 0 to 24 Hours Post Dose Measured on Day 30 (AUC (0-24))
Description: as for outcome 8
Time Frame: T0 (predose), T1hour (hr), T2hr, T4hr, T6 hr, T8 hr, T10hr, T12hr, T16hr, T24hr, T32hr, T36hr, T48hr, T72hr (post dose)
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Differin® Gel, 0.3% | Differin® Gel, 0.1%
Number analyzed (Participants) | 25 | 25
ng*h/mL | 2.64 (1.66) | 0.42 (1.03)

ADVERSE EVENTS:
Arm/Group | Differin® Gel, 0.3% | Differin® Gel, 0.1%
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 3/26 | 2/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Differin® Gel, 0.3% (N=26) | Differin® Gel, 0.1% (N=25)
Joint sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No